CLINICAL TRIAL: NCT05684081
Title: Effectiveness of Mobile Money Payments to Vaccination Campaign Health Care Workers on Polio Vaccination Campaign Coverage and Quality: a Cluster Randomized Controlled Trial
Brief Title: Effect of Digital Payment to Campaign Health Workers on Vaccination Coverage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MaKSPH_BMGF_INV03047_2022
Record Dates: First submitted 2022-11-17; First posted 2023-01-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Polio
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: The intervention consists of direct cash payment to vaccination campaign health workers using government of Uganda Ecash platform on IFMIS
Masking Description: This is an unblinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): Refers to the intervention arm i.e. ECASH payment of health workers
  Interventions: Behavioral: Digital payment
- CONTROL (No Intervention): Refers to status Quo or no intervention i.e. payment using cash

INTERVENTIONS:
Behavioral: Digital payment — The proposed intervention is designed to support the implementation of polio campaigns through digital payments
  Arms: INTERVENTION

SUMMARY:
Introduction:

Good quality OPV campaigns can interrupt and possibly prevent transmission of the polio virus. Health care worker performance and motivation are prerequisites for the success of such campaigns. Complete, transparent and timely payments are, in turn, prerequisites for the sustenance of health care worker motivation and thereby efforts. To date, most such health care workers have been paid in cash, with chronic payment issues that have negatively affected campaign quality and vaccination coverage. Cash-based payments are often plagued with multiple delays in funds disbursements, cash leakages, and a lack of accountability and financial transparency. These difficulties have prompted a transition to digitized payments that are perceived to be faster, more convenient, traceable, reliable, easier and more reasonable to set up. The roll-out phase of these digital payment interventions has not been quantitatively evaluated and the effect of digital payments on the motivation, satisfaction and performance of health workers is not known. Therefore, this study will compare digitized payment of polio vaccination campaign health care workers with cash-based payment with regards to health care worker motivation, satisfaction and performance. Findings from this study may inform the operationalization of digital financial systems, and the transition towards cross-campaign digital payments.

Primary Objectives:

1. To compare the motivation, satisfaction and performance of vaccination health care workers in areas where they are paid using mobile money versus in cash,
2. To explore how gender norms and relations influence health workers' response to payment systems (mobile money versus cash payments) and how these affect the health workers' performance and motivation in polio vaccination campaigns and

Secondary objectives:

1. To compare vaccination campaign quality in areas where health care workers are paid using mobile money versus in cash
2. To compare vaccination coverage in areas where campaign health care workers are paid using mobile money versus in cash.
3. To estimate the incremental cost of the intervention.

Methods:

This will be a mixed methods study including a cluster-randomized controlled implementation trial and a qualitative study. A total of 60 districts be randomized to implement either a digital payment system for polio campaign vaccinators during the polio campaign or the traditional cash-based payment system.

DETAILED DESCRIPTION:
Problem statement and justification

A motivated health workforce is essential for the success of critical health campaigns and programmes such as the recently concluded and upcoming polio campaigns. This is even more critical particularly in periods during and following disruptions in health services such as the Covid-19 pandemic and the resultant restrictions. Remuneration, which has been traditionally cash based is a key factor for health care worker motivation, satisfaction and performance. However, traditional cash-based modes of payment are fraught with numerous problems like delays in funds requisitions and disbursements, cash leakages, exposure to risk of theft while in transit, and a lack of accountability data and financial transparency. These chronic problems associated with cash-based payments have led to a gradual transition to digital (mobile money) payments in several countries including Uganda. While digital payments are seen as fast, convenient, traceable, reliable, and easy to set up, they are not themselves free of challenges. Also, their effect on health outcomes has not been evaluated with robust scientific methods.

Few studies have particularly paid attention to the role of digital payments in influencing gender relations (power relations, access to resources and gender roles) and also how gender relations affect the adoption and use of digital payments particularly in relation to health worker's motivation and performance that is essential for increasing coverage and quality of vaccination campaigns. Furthermore, the investigators are cognizant of the intersections between gender and other social identities of both female and male health workers such as gender, age, education, cadre of health worker, income bracket, location, disability, ethnicity) that could have a bearing on how they interact and respond to digital payments-and their implications on the motivation and performance of health workers.

This study therefore, will evaluate an intervention that seeks solutions to the current challenges faced by payment systems by providing a verified national database of health care workers and processing payments directly to those health care workers digitally, through mobile money platforms. Set within the context of the upcoming polio vaccination campaign, this study will examine the effect of this intervention on health outcomes such as polio vaccination coverage as well as health worker related outcomes like motivation, satisfaction and performance. This study will also examine the effect of gender norms/gender relations on health workers' response to payment systems employed during polio vaccination. While maintaining Uganda free of polio is in itself a very important goal, lessons learned from this cluster randomized implementation trial can be extended to other health campaigns and programmes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and above
2. History of participation in the most recent polio vaccination campaign in Uganda
3. Member of the district leadership team

Exclusion Criteria:

1) Non-consenting adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Vaccination campaign health care worker motivation, performance and satisfaction based on self reports on a scale of 1-5 | At least one week post payment of immunization health workers
  Assessing the health workers motivation, performance and satisfaction based on self report on a scale of 1-5.

SECONDARY OUTCOMES:
Vaccination coverage | At least one week post payment of immunization health workers
  Proportion of children 0-59 vaccinated against polio during the campaign

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Nankabirwa, PhD, Principal Investigator — Makerere University
Locations (1):
- Ministry of Health Facilities in 54 districts/municipalities in Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waiswa P, McConnell M, Aweko J, Mukuye DD, Opio C, Ashaba MS, Bakainaga A, Ekirapa-Kiracho E. The effect of supporting districts to operationalise digital payments for vaccination campaign workers: a cluster randomised controlled trial during the 2022 polio vaccination campaign in Uganda. BMJ Glob Health. 2025 Sep 10;10(Suppl 4):e016666. doi: 10.1136/bmjgh-2024-016666. PMID 40935396